CLINICAL TRIAL: NCT06879990
Title: The Role of Retrograde Saline Irrigation Through Double Lumen Ureteric Catheter During Supine Mini-percutanous Nephrolithotomy for Renal Stones Extraction:a Prospective Controlled Trial
Brief Title: Retrograde Saline Irrigation During Supine Mini Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Elsayed Abdelhalim Elsayed, assistant lecturer, urology department, Kafrelsheikh university,Msc, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 36264PR17/1/23
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Renal Stone; Supine Mini Percutaneous Nephrolithotomy
Keywords: Supine
MeSH Terms: conditions — Nephrolithiasis; Deception

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine mini percutaneous nephrolithotomy with irrigation (Experimental)
  Interventions: Behavioral: Retrograde normal saline irrigation
- Supine mini percutaneous nephrolithotomy without irrigation (Experimental)
  Interventions: Behavioral: Without Retrograde normal saline irrigation

INTERVENTIONS:
Behavioral: Retrograde normal saline irrigation — Retrograde normal saline irrigation during supine Mini percutaneous nephrolithotomy
  Arms: Supine mini percutaneous nephrolithotomy with irrigation
Behavioral: Without Retrograde normal saline irrigation — Without Retrograde normal saline irrigation during supine Mini percutaneous nephrolithotomy
  Arms: Supine mini percutaneous nephrolithotomy without irrigation

SUMMARY:
This minimally invasive surgery allows us to remove kidney stones through tiny incisions and provides patients with quicker and smoother recoveries

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* renal stones

Exclusion Criteria:

* age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Stone free rate | two weeks from primary procedure
  No stone residual fragments

SECONDARY OUTCOMES:
Assess operative time | During procedure
  Assess operative time in minutes
Post operative complication | Up to 48 hours
  Complication may occur post operative like fever , sever pain

CONTACTS AND LOCATIONS:
Locations (1):
- Elsayed Abdelhalim, Kafr ash Shaykh, State, Egypt